CLINICAL TRIAL: NCT02728154
Title: Characterize the Gut Microbiota in Subjects With Heart Failure and Pre-heart Failure With Preserved Ejection Fraction
Brief Title: The Role of Gut Microbiota in Heart Failure and Pre-Heart Failure With Preserved Ejection Fraction
Status: Withdrawn | Type: Observational
Why Stopped: No study participants enrolled
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600380 - N
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: pre-clinical diastolic dysfunction (pre-HFpEF)
MeSH Terms: conditions — Heart Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal control: The subjects in the normal heart function group will provide a blood sample and stool sample.
  Interventions: Other: Blood Sample; Other: Stool Sample
- heart failure: The subjects in history of heart failure group will provide a blood sample and stool sample.
  Interventions: Other: Blood Sample; Other: Stool Sample
- pre-HFpEF: The subjects in history of diastolic dysfunction but not had heart failure clinical presentations group will provide a blood sample and stool sample.
  Interventions: Other: Blood Sample; Other: Stool Sample

INTERVENTIONS:
Other: Blood Sample — One tablespoon of blood will be drawn once during the study.
Other: Stool Sample — One stool sample will be collected.

SUMMARY:
Gut microbiota play an important role in normal cardiovascular function and pathophysiology of cardiovascular diseases. Patients with heart failure (HF) have substantial hemodynamic changes which lead to intestinal hypoperfusion and congestion and eventually change gut morphology, permeability, function and composition of gut microbiota and cause translocation of microbial and endotoxins into the blood stream. Additionally, metabolites derived from gut microbiota modulate the pathophysiology of HF. Patients with HF have intestinal overgrowth of pathogenic bacteria and increased gut permeability. Accumulating evidence demonstrates that antibiotic treatment benefits patients with acute coronary syndromes and reduces the incidence of ischemic cardiovascular events. Taking the strong association of gut microbiota with HF into account, it is reasonable to speculate that gut microbiota could contribute to the progression of pre-HF with preserved ejection fraction (pre-HFpEF) to HF with preserved ejection fraction (HFpEF). Pre-HFpEF remains poorly understood, yet has high prevalence and a significantly high risk for death in comparison to patient without pre-HFpEF. We hypothesize that altered gut microbiota is involved in the initiation and establishment of HF and pre-HFpEF.

DETAILED DESCRIPTION:
The research study will initially enroll 50 subjects without HF as normal controls,120 subjects with history of HF and 50 subjects with pre-HFpEF to characterize gut microbiota. The subjects will provide blood samples and a stool sample.

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to provide consent
* Control subjects with normal heart function
* Subjects with history of HF
* Subjects with impaired ventricular relaxation and/or elevated left ventricular end diastolic pressure measured by echocardiography and/or catheterization, yet has not had HF clinical presentations

Exclusion Criteria:

* intestinal surgery,
* inflammatory bowel disease,
* celiac disease,
* lactose intolerance,
* chronic pancreatitis or
* other malabsorption disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consenting participants who have normal, diastolic dysfunction or heart failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2025-06-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Stool sample for fecal microbiota between the groups | Day 1
  Stool samples will be collected to compare the fecal microbiota of subjects with normal, diastolic heart dysfunction before heart failure developed and heart failure.

SECONDARY OUTCOMES:
Blood samples for inflammatory cytokines between the groups | Day 1
  Blood samples will be used to compare difference in inflammatory cytokines including Interleukin-1 (IL-1), 6, 17 between groups using ELISA kits.
Blood samples for SAA between the groups | Day 1
  Blood samples will be used to compare difference in serum amyloid (SAA) a between groups using ELISA kits.
Blood samples for inflammatory cells between the groups | Day 1
  Blood samples will be used for difference in progenitor/inflammatory cells between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- Cardiovascular Clinic at UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided